CLINICAL TRIAL: NCT04340427
Title: A Phase I Study of TQB3455 Tablets in Subjects With Advanced Malignancies
Brief Title: A Study of TQB3455 Tablets in Subjects With Advanced Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3455-I-02
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3455 Tablets (Experimental): TQB3455 Tablet administered orally once. Then TQB3455 Tablet administered orally, once daily in 28-day cycle after 7 days of first administration.
  Interventions: Drug: TQB3455

INTERVENTIONS:
Drug: TQB3455 — TQB3455 tablets is a small molecule oral drug inhibiting IDH2 mutation.

SUMMARY:
This is a open-label, multicenter, phase I study to evaluate tolerance and pharmacokinetics of TQB3455 tablets in subjects with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥ 18 years old； Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2; Life expectancy ≥12 weeks.

  2. Has IDH2 gene mutation will be selected preferentially. 3. The toxicity of radiotherapy or other antitumor therapy should return to grade 1.

  4. No pregnant or lactating women, all the participants should use contraceptives.

  5. Understood and signed an informed consent form. 6. Advanced/metastatic solid tumors or refractory/recurrent acute myeloid leukemia.

  7. At least one measurable lesion for solid tumors. 8. Adequate organ system function.

Exclusion Criteria:

* 1.Relapsed after bone marrow transplantation. 2.Has received systemic antitumor therapy or radiation therapy within 3 weeks before the first dose.

  3.Has participated in other clinical trial within four weeks before the first dose.

  4.Has multiple factors affecting oral medication. 5.Has uncontrolled, active systemic fungal, bacterial, or viral infections. 6.Poorly controlled hypertension. 7.Has serious cardiovascular disease. 8.Has drug abuse history that unable to abstain from or mental disorders. 9.Has active hepatitis B or C. 10.Have a history of immunodeficiency. 11.According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

  12.Has central nervous system metastasis with the exception of glioma subjects. 13.Has severe life-threatening complication of leukemia, such as uncontrolled bleeding, hypoxia or shock pneumonia, and disseminated intravascular coagulation.

  14.Has central nervous system leukemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days
  Subjects appear the toxic reaction relate to the drug after treatment within 28 days.

SECONDARY OUTCOMES:
Cmax | Hour 0, 1, 2, 3, 5, 8, 10, 12, 24, 48, 72, 96, 120, 144 hours post-dose on single dose; Hour 0 of day 8, day 15, day22 on multiple dose and hour 0, 1, 2, 3, 5, 8, 10, 12, 24 hours post-dose on multiple dose of day 28.
  Cmax is the maximum plasma concentration of TQB3455 or metabolite(s).
Tmax | Hour 0, 1, 2, 3, 5, 8, 10, 12, 24, 48, 72, 96, 120, 144 hours post-dose on single dose; Hour 0 of day 8,day 15,day22 on multiple dose and hour 0, 1, 2, 3, 5, 8, 10, 12, 24 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3455 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 1, 2, 3, 5, 8, 10, 12, 24, 48, 72, 96, 120, 144 hours post-dose on single dose; Hour 0 of day 8,day 15,day22 on multiple dose and hour 0, 1, 2, 3, 5, 8, 10, 12, 24 hours post-dose on multiple dose of day 28.
  To characterize the pharmacokinetics of TQB3455 by assessment of area under the plasma concentration time curve from zero to infinity.
α-Hydroxyglutaric acid (2-HG) | Day 1, Day 8 and Day 15 pre-dose on cycle 1; Day1, Day15 pre-dose on cycle 2 and cycle 3; Day 1 pre-dose on multiple dose from cycle 4 to cycle 8. Each cycle is 28 days.
  The concentration of 2-HG.

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China